CLINICAL TRIAL: NCT00456196
Title: Epidemiology of Venous Thromboembolism: Analyses and Publications From the DVT FREE Database
Brief Title: Epidemiology of Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Samuel Z. Goldhaber, MD, Brigham and Women's Hospital
Other Study IDs: 2006-P-000820
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Venous Thromboembolism; Pulmonary Embolism; Cancer; Deep Vein Thrombosis; COPD
Keywords: COPD; Thrombosis; Cancer; Renal; Elderly; Surgery; Orthopedic Surgery; Medically Ill; Deep Vein Thrombosis; Pulmonary Embolism; Anticoagulation
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism; Neoplasms; Venous Thrombosis; Pulmonary Disease, Chronic Obstructive; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
More than 5 years ago the DVT FREE Registry was conceived. Its database consists of 5,451 ultrasound-confirmed DVT patients from 183 institutions. This database is rich in information of critical importance to health care providers. The information contained within the database will be revisited to provide more detailed analyses which will be used for risk factor assessment and for decision-making regarding the implementation of VTE Prophylaxis.

DETAILED DESCRIPTION:
BACKGROUND:

The Venous Thromboembolism (VTE) Research Group has explored and studied the epidemiology of DVT and pulmonary embolism (PE) for more than 2 decades. The earliest analyses were done with the database from the Framingham Heart Study. Subsequent analyses were undertaken using the Nurses' Health Study.

More than 5 years ago the DVT FREE Registry was conceived. The concept was to accrue broad representation of patients with ultrasound-confirmed DVT throughout the US.

The Principal Investigator began initial work on this project by developing the case report form (CRF) with Co-Investigators. After the CRF was piloted and finalized, centers were recruited for participation. The enthusiasm in response to DVT FREE was overwhelming. The initial investigators meetings were conducted by videoconference shortly after September 11, 2001. Accrual of patients occurred much more rapidly than projected. Within 6 months, 5,451 patients were enrolled with ultrasound-confirmed DVT at 183 participating institutions.

Dr. Samuel Z. Goldhaber chaired the Publications Committee. The Master Paper was published in January 2004. 3 manuscripts on subgroups and 3 manuscripts on special populations were subsequently published under Dr. Goldhaber's supervision. The subgroup papers studied upper extremity DVT, the relationship between DVT and symptomatic DVT and PE, and predictors of massive DVT. The special populations papers studied gender differences in receiving prophylaxis, utilization of vena cava filters, and pregnancy.

Though the publication record is impressive in scope, much work remains to be done. The database is rich in information of critical importance to health care providers. The information contained within the database should be analyzed to provide more detailed analyses which will be used for risk factor assessment and for decision-making regarding the implementation of VTE prophylaxis.

For the current DVT FREE publication project, we will use the database to analyze findings that will yield 8 publications in special populations: 1) medically ill hospitalized patients, 2) cancer patients, 3) nonorthopedic general surgery patients, 4) orthopedic surgery patients, 5) long-haul travel patients, 6) COPD Patients, 7) Renal Patients, and 8) Elderly Patients.

PROJECT DESCRIPTION:

1. Medically Ill Hospitalized Patients:

   Medically ill hospitalized patients are the most important subgroup to study. These patients often do not receive guideline-recommended prophylaxis. We believe that medically ill hospitalized patients are underserved.

   For this DVT FREE publication, we will exclude all patients who had surgery within the past 3 months. We will also exclude women who were pregnant or postpartum. All other patients will be included in these analyses. They will be stratified according to age, height, weight, body mass index (BMI), gender, and whether they received prophylaxis.
2. Cancer Patients:

   Cancer patients have received increasing attention because of the relationship between cancer and DVT. For example, the National Comprehensive Cancer Network (NCCN) organized a special committee to write consensus guidelines for prevention and treatment of DVT in this patient population.

   For this DVT FREE publication, we will include all patients with cancer. We will also include whether the cancer was active and whether the patient is receiving ongoing radiation therapy or chemotherapy. These cancer patients will be stratified according to age, height, weight, BMI, gender, and whether they received prophylaxis.
3. Nonorthopedic General Surgery Patients:

   For this DVT FREE publication, we will include all nonorthopedic general surgery patients. These patients will have undergone surgery within the 3 months prior to DVT. We will also explore the type of surgery (excluding orthopedic surgery) and type of anesthetic that was used. These patients will be stratified according to age, height, weight, BMI, gender, and whether they received prophylaxis.
4. Orthopedic Surgery Patients:

   For this DVT FREE publication, we will include all orthopedic surgery patients. We will also include patients who suffered hip fracture, pelvic fracture, upper extremity fracture, lower extremity fracture, or other fracture within 30 days prior to enrollment. We will also include patients with major trauma to the spine, pelvis, or upper or lower extremities. These patients will be stratified according to age, height, weight, BMI, gender, and whether they received prophylaxis.
5. Congestive Heart Failure (CHF)
6. COPD Patients:

   For this DVT FREE publication, we will include all patients with COPD. These patients will be stratified according to age, height, weight, BMI, gender, and whether they received prophylaxis.
7. Renal Patients:

   For this DVT FREE publication, we will include all renal patients. These patients will be stratified according to age, height, weight, BMI, gender, and whether they received prophylaxis.
8. Elderly Patients:

For this DVT FREE publication, we will include all elderly patients. For this study we will define elderly as 70 years of age or older. These patients will be stratified according to age, height, weight, BMI, gender, and whether they received prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound-confirmed DVT patients from 183 institutions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the DVT FREE study with ultrasound-confirmed deep vein thrombosis
Sampling Method: Non-Probability Sample
Enrollment: 5451 (Actual)
Dates: Start 2006-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Z. Goldhaber, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Joffe HV, Kucher N, Tapson VF, Goldhaber SZ; Deep Vein Thrombosis (DVT) FREE Steering Committee. Upper-extremity deep vein thrombosis: a prospective registry of 592 patients. Circulation. 2004 Sep 21;110(12):1605-11. doi: 10.1161/01.CIR.0000142289.94369.D7. Epub 2004 Sep 7. PMID 15353493
- [Background] Kucher N, Tapson VF, Goldhaber SZ; DVT FREE Steering Committee. Risk factors associated with symptomatic pulmonary embolism in a large cohort of deep vein thrombosis patients. Thromb Haemost. 2005 Mar;93(3):494-8. doi: 10.1160/TH04-09-0587. PMID 15735800
- [Background] Joffe HV, Kucher N, Tapson VF, Goldhaber SZ. Few predictors of massive deep vein thrombosis. Thromb Haemost. 2005 Nov;94(5):986-90. doi: 10.1160/TH05-05-0314. PMID 16363241
- [Result] Goldhaber SZ, Tapson VF; DVT FREE Steering Committee. A prospective registry of 5,451 patients with ultrasound-confirmed deep vein thrombosis. Am J Cardiol. 2004 Jan 15;93(2):259-62. doi: 10.1016/j.amjcard.2003.09.057. PMID 14715365
- See also: North American Thrombosis Forum — http://www.NATFonline.org